CLINICAL TRIAL: NCT05893238
Title: Human Follicular Fluid Markers and Reproductive Outcomes in IVF: Relevant Factors for the Oocyte's Developmental Potential
Brief Title: Human Follicular Fluid Markers and Reproductive Outcomes in IVF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Janna Pape (Other)
Responsible Party: Sponsor-Investigator, Janna Pape, Principal Investigator, Senior doctor, Janna Pape (MD), Universitätsklinik fur Frauenheilkunde, Inselspital Bern
Organization: Universitätsklinik fur Frauenheilkunde, Inselspital Bern (Other)
Other Study IDs: KEK Bern 2022-00944
Record Dates: First submitted 2023-05-18; First posted 2023-06-07 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-05

CONDITIONS: IVF; Infertility
Keywords: Natural IVF; Follicular Fluid; Oxidation-reduction potential; Gonadotrophin; Lifestyle
MeSH Terms: conditions — Infertility | interventions — Blood Specimen Collection; Congresses as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Follicular fluid; serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- In Vitro Fertilisation (IVF)-Patients without hormonal stimulation (Natural cycle IVF): Natural cycle IVF
  Interventions: Procedure: Natural cycle In Vitro Fertilisation (IVF); Diagnostic Test: Blood samples for analysis; Diagnostic Test: Follicular fluid for analysis; Diagnostic Test: Sperm samples for analysis
- In Vitro Fertilisation (IVF)-Patients with hormonal stimulation (conventional IVF): conventional IVF
  Interventions: Diagnostic Test: Blood samples for analysis; Diagnostic Test: Follicular fluid for analysis; Diagnostic Test: Sperm samples for analysis; Procedure: Conventional In Vitro Fertilisation (IVF)

INTERVENTIONS:
Procedure: Natural cycle In Vitro Fertilisation (IVF) — In Vitro Fertilisation (IVF) without hormonal stimulation
  Groups: In Vitro Fertilisation (IVF)-Patients without hormonal stimulation (Natural cycle IVF)
Diagnostic Test: Blood samples for analysis — Test hormone levels in serum
Diagnostic Test: Follicular fluid for analysis — Test hormone levels in follicular fluid Test Oxidation-reduction potential
Diagnostic Test: Sperm samples for analysis — Oxidation-reduction potential
Procedure: Conventional In Vitro Fertilisation (IVF) — In Vitro Fertilisation (IVF) with conventional hormonal stimulation
  Groups: In Vitro Fertilisation (IVF)-Patients with hormonal stimulation (conventional IVF)

SUMMARY:
The goal of this observational study is to understand the processes in the growing follicles development in more detail and to improve In Vitro Fertilisation (IVF) treatments. This involves measuring laboratory values in the blood, in the follicular fluid of the woman and in the sperm of the man as well as questionnaires concerning lifestyle factors. These values are then linked to the success of the fertility treatment to find out which of these values increase the success of the IVF treatment.

Furthermore, the investigators want to investigate if there are differences between IVF treatments with or without hormonal stimulation of the ovaries.

DETAILED DESCRIPTION:
This is a one-site prospective exploratory study at the University Clinic for Gynaecological Endocrinology and Reproductive Medicine in Bern. Data of influencing factors on IVF success in women and men will be collected in two types of IVF treatment, i.e. with or without hormonal stimulation of the ovaries.

The investigators want to

* compare the follicular fluid values between the two IVF treatment groups.
* assess the associations and predictive power of follicular fluid / blood and sperm parameters for success of the IVF treatment.
* compare the IVF success in the two treatment groups. The study aims to enrol approximately 200 couples. The data will be collected by the physicians and added to the REDcap study registry. Access to the total data set is only permitted for the principal investigator.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate
* Written consent
* Couples undergoing In Vitro Fertilisation (natural cycle or conventional IVF)

Exclusion Criteria:

* Not willing to participate
* Missing consent
* Female of the couple does not want to participate or missing consent
* Language barrier
* Medical freezing
* Social freezing
* Thawed cycles
* Genetic disorders
* Preimplantation genetic testing (PGT)
* Medication for chronic condition
* Surgery in the last 4 weeks
* Significant trauma in the last 90 days
* Severe reduced sperm quality
* Kryosperm
* Poor responder or expected poor response

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients aiming to do In Vitro Fertilisation with fresh embryo transfer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Blastocyst rate per oocyte | 5 days after fertilization
  Number of blastocysts out of fertilized oocytes observed 5 days after fertilization

SECONDARY OUTCOMES:
Number of mature oocytes | 4-6 hours after punction
  Number of mature oocytes from punctured follicles
Cleavage rate per oocyte | 2 days after fertilization
  Number of cleavage embryos out of fertilized oocytes observed 2 days after fertilization
Morphologic evaluation of blastocyst | 5 days after fertilization
  Morphologic evaluation according to the Gardner score (Gardner and Schoolcraft, 1999)
Implantation rate | 10-12 days after embryo transfer
  Endocrine pregnancy by measuring hCG in blood sample on day 10-12 after embryo transfer
Clinical pregnancy rate | 5 weeks after embryo transfer
  Clinical pregnancy confirmed by ultrasound, 5 weeks after embryo transfer.
Live birth rate | 9 months after embryo transfer
  Birth of a living baby nine months after embryo transfer

CONTACTS AND LOCATIONS:
Locations (1):
- Inselspital Bern, Frauenklinik, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No